CLINICAL TRIAL: NCT00959361
Title: Evaluation of Effectiveness of Pharmaceutical Care on the Adherence of HIV-Positive Patients to Antiretroviral Therapy - Randomized Clinical Trial
Brief Title: Evaluation of Effectiveness of Pharmaceutical Care on the Adherence of HIV-Positive Patients to Antiretroviral Therapy
Acronym: PC-HIV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Collaborators: Federal University of Rio Grande do Sul (Other)
Responsible Party: Marysabel Pinto Telis Silveira, Universidade Católica de Pelotas
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2003164
Record Dates: First submitted 2009-08-13; First posted 2009-08-14 (Estimated); Last update posted 2009-09-29 (Estimated); Status verified 2009-08

CONDITIONS: HIV; HIV Infections
Keywords: patient compliance; guidelines adherence; advance directive adherence; treatment refusal; directly observed therapy; anti-retroviral agents; HIV seropositivity; HIV infections; HIV; pharmaceutical services; HIV-positives patients; treatment experienced
MeSH Terms: conditions — HIV Infections; Patient Compliance; Treatment Refusal; Directly Observed Therapy; HIV Seropositivity | interventions — Pharmaceutical Services

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- pharmaceutical care (Experimental): consultation with the pharmacists
  Interventions: Behavioral: pharmaceutical care
- control (No Intervention): usual care without consultation with the pharmacists

INTERVENTIONS:
Behavioral: pharmaceutical care — consultation with the pharmacists and usual care
  Other Names: pharmaceutical attention; DADER method
  Arms: pharmaceutical care

SUMMARY:
INTRODUCTION: Studies prove that the pharmaceutical care (PC) increases the adherence to the antiretroviral; thus, they increase the undetectable viral load. The viral load diminishes, and the prevalence of undetectable viral load increases, as the levels of adherence to the treatment increase, being in general necessary high adhesion to reach the effectiveness therapeutic. Increasing the adherence levels, it increases the surviving chances and quality of life and diminishes the transmission risks. Studies demonstrate that the self-effectiveness expectation to use the medication correctly is the main predictor of adherence, and that the more complex the therapeutic regimen is, and the perception of side effects, the smaller the adherence is, highlighting the importance of preventing, identifying and solving the problems during the treatment with antiretroviral, problems related to the medication (PRM) through the PC.

OBJECTIVES: To evaluate the effectiveness of the PC on the adherence of HIV-patients to the antiretroviral therapy, identify, prevent and solve PRMs during the treatment.

METHODOLOGY: One-side randomized clinical trail controlled by non-intervention in parallel. 332 patients randomized are included in the control and intervention groups (PC). Questionnaires will be applied: sociodemographic, adherence to the antiretroviral through self-report, smoke, BECK (depression), CAGE (problems related with alcohol consumption) of self-effectiveness, expectation of results and social support. Each 4 months measure of viral load and CD4 will be carried out. The ones from the PC group will receive a card with information about the medication and all the medicines will be identified by different colors. The follow-up will last one year according to the instructions of DADER program.

DETAILED DESCRIPTION:
Election of the sample: 332 will be selected consecutively patients registered in the SAE-Pelotas

GENERAL OBJECTIVE To evaluate the effectiveness of Pharmaceutical Care on the adherence to the antiretroviral therapy in HIV- positive patients.

PRIMARY OBJECTIVE The relative risk for adherence to the antiretroviral treatment among HIV-positive patients who receive Pharmaceutical Care and the ones that do not receive Pharmaceutical Care is different of 1.

SECONDARY OBJECTIVE The relative risk for undetectable viral load among HIV-positive patients that receive Pharmaceutical Care and the ones that do not receive Pharmaceutical Care is different of 1.

ELIGIBILITY:
Inclusion Criteria:

* patients registered in the SAE-Pelotas
* adults (older 18 years)
* inhabitants of the urban zone of Pelotas
* not pregnant
* in use of antiretroviral treatment
* independent of the time of treatment
* accept to participate in the research through the signature of a written informed consent

The enclosed patients will be randomized through program computerized for the group of pharmaceutical care or control group.

Exclusion Criteria:

* non signature of a written informed consent
* incapacity to answer to the instruments of data collection
* inhabitants are of the urban zone of Pelotas
* patients who could not be followed by 12 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 332 (Actual)
Dates: Start 2006-06; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Relative risk for adherence to the antiretroviral treatment among HIV-positive patients who receive Pharmaceutical Care and the ones that do not receive Pharmaceutical | one year

CONTACTS AND LOCATIONS:
Overall Officials: LEILA B MOREIRA, DR, Principal Investigator — Hospital de Clínicas de Porto Alegre
Locations (1):
- Hospital de Clinicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil